CLINICAL TRIAL: NCT05870969
Title: Exploration of A Holistic Management Procedure for Liver Cancer Surveillance in Improving Liver Cancer's Early Diagnosis Efficacy in Chinese Population: Single-Center, Prospective, Observational Real-world Study in EASTERN China
Brief Title: Digitalized Surveillance Management for Liver Cancer Risk Population in Improving Eearly Diagnosis Efficancy in Chinese Population (dSEARCH)
Acronym: dSEARCH
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Qing XIe, Director of Department of Infectious Diseases, Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Ruijin Hospital
Other Study IDs: dSEARCH
Record Dates: First submitted 2023-05-13; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma, Hepatocellular; Hepatitis C, Chronic; Hepatitis B, Chronic; Cirrhosis, Liver; Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis C, Chronic; Hepatitis B, Chronic; Liver Cirrhosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with very high risk for HCC according local guideline
  Interventions: Behavioral: Liver cancer surveillance every 3 months
- Patients with high risk for HCC according local guideline
  Interventions: Behavioral: Liver cancer surveillance every 3 months
- Patients with medium risk for HCC according local guideline
  Interventions: Behavioral: Liver cancer surveillance every 6 months
- Patients with low risk for HCC according local guideline
  Interventions: Behavioral: Liver cancer surveillance annually

INTERVENTIONS:
Behavioral: Liver cancer surveillance every 3 months — Follow up every 3 months for liver cancer surveillance, including but not limited to serum AFP test and ultrasound exam
  Groups: Patients with high risk for HCC according local guideline; Patients with very high risk for HCC according local guideline
Behavioral: Liver cancer surveillance every 6 months — Follow up every 6 months for liver cancer surveillance, including but not limited to serum AFP test and ultrasound exam
  Groups: Patients with medium risk for HCC according local guideline
Behavioral: Liver cancer surveillance annually — Follow up annually for liver cancer surveillance, including but not limited to serum AFP test and ultrasound exam
  Groups: Patients with low risk for HCC according local guideline

SUMMARY:
The goal of this study is to evaluate whether the standardized liver cancer risk stratification management can effectively improve the early diagnosis rate of liver cancer in the targeted risk population in China.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation in the clinical study; fully informed about the study and signed informed consent, willing to follow and capable of completing all trial procedures[17]
2. Age: 18 to 75 years old (including the cut-offs)
3. Subjects must meet at least one of the following criteria for enrollment.

   1. Patients diagnosed with chronic hepatitis B in hospital or out of hospital: persistent positive hepatitis B surface antigen (HBsAg) for 6 months or more
   2. Patients diagnosed with hepatitis C in hospital or out of hospital
   3. Patients diagnosed with cirrhosis in hospital or out of hospital who meet at least one of the following criteria.

      1. Liver biopsy showing cirrhosis (Ishak score ≥5 or Metavir score = 4);
      2. Liver stiffness measurement (LSM) using FibroScan® (Echosens™, Paris, France) ≥12.0 kPa when TB was normal and ALT ≤ 40 IU/mL, or LSM ≥ 17.0 kPa when TB was normal and ALT < 200 IU/mL;
      3. Abdominal imaging results showing characteristic of cirrhosis (results showing coarse liver echotexture or nodular, parenchymal, or morphological abnormalities and signs of gastroesophageal varices);
      4. APRI ≥ 2.0;
      5. FIB-4 ≥ 3.25
   4. Patients diagnosed with metabolic dysfunction-associated fatty liver disease (MAFLD) in hospital or out of hospital who have a liver fibrosis score of F3 or higher according to transient elastography, i.e., FibroScan® Liver Stiffness Measurement (LSM) ≥ 10 kPa or the corresponding FibroTouch® measurement threshold[18].

      * MAFLD diagnosis requires diagnosis of >5% fat accumulation in liver through either FibroScan® CAP measurements, or similar parameter, or liver biopsy, and in combination with one of the following three conditions: overweight/obesity (BMI >23 kg/m2), type 2 diabetes, or metabolic dysfunction.
   5. Patients diagnosed with MAFLD combined with abnormal glucose metabolism[19]

      * Abnormal glucose metabolism is defined as type 2 diabetes, or prediabetes, i.e. fasting blood glucose 5.6-6.9 mmol/L, or 2h postprandial blood glucose 7.8-11.0 mmol/L, or glycated hemoglobin 5.7%-6.4%
   6. Subjects with a family history of liver cancer in their first-degree biological relatives.

Exclusion Criteria:

Patients meeting any of the following criteria will be excluded from the study:

1. Age <18 years or >75 years
2. Patients who have been diagnosed with liver cancer before enrollment
3. Patients with severe mental illness or cognitive impairment
4. Patients who are pregnant or lactating, or preparing to become pregnant
5. Patients who have participated in other clinical trials or are participating in other clinical trials within 3 months prior to initiation of study treatment
6. According to the doctor's judgment, the possibility of the subject being included is low (including inability to understand the project requirements , poor compliance, infirmity, inability to ensure that the protocol can be implemented as required, etc.), or the doctor determines that the subject has any other factors that are not suitable for this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study mainly includes the following risk groups of liver cancer: patients with chronic hepatitis B, patients with hepatitis C, patients with liver cirrhosis, patients with metabolic dysfunction-associated fatty liver disease (MAFLD) with a liver fibrosis index F3 or above, MAFLD patients combined with abnormal glucose metabolism, and people with a family history of liver cancer in their first-degree biological relatives.
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Early diagnosis rate of HCC patients | Follow up up to three years for HCC occurance.
  The proportion of patients who are first diagnosed with HCC at early stage to all the patients diagnosed as liver cancer in the study, from the start of the study to the completion of follow-up. Early diagnosis is defined as the patient with stage CNLC Ia, Ib and IIa.

SECONDARY OUTCOMES:
Proportion of subjects with regular follow-up | Four years collectively after the study started
  Regular follow-up is defined as the average difference between the actual treatment time and the theoretical treatment time equal or less than 1/3
  * Actual visit interval: actual visit date - previous visit date ② Theoretical visit interval: theoretical visit date (the date that physician advise to return to hospital for visit) - previous visit date ③ Follow-up compliance = (②-①)/② ④ Patient with regular follow-up is defined as the patient whose mean follow-up compliance is equal to, or less than 1/3
    * The compliance of the study is defined as the proportion of subjects with regular follow-up to all subjects in the study.
The distribution of risk stratification of liver cancer in subjects at initial screening | Initial screening after enrollment
  The proportion of very high-risk, high-risk, medium-risk, and low-risk subjects to the whole subject population
The distribution of risk stratification of liver cancer in subjects at the last follow-up visit or at the time of diagnosis of liver cancer | Last follow-up visit or at the time of diagnosis of liver cancer up to three years of follow-up
  The proportion of very high-risk, high-risk, medium-risk and low-risk subjects to the whole subject population
Pooled 3-year cumulative incidence of liver cancer | Follow up up to 3 years
The early diagnosis rate of liver cancer in each subject category according to the risk stratification at initial screening | Initial screening after enrollment
  The early diagnosis rate of liver cancer of subjects with very high-risk, high-risk, medium-risk, and low-risk at initial screening, respectively
The 3-year cumulative incidence of liver cancer in each subject category according to the risk stratification at the time of initial diagnosis | Four years collectively after the study started
  The 3-year cumulative incidence of liver cancer for subjects with very high-risk, high-risk, medium-risk, and low-risk, respectively

OTHER OUTCOMES:
The number of patients first diagnosed with liver cancer and the annual incidence rate | Four years collectively after the study started
The number of patients first diagnosed with liver cancer and the annual incidence rate within each risk category | Four years collectively after the study started
The distribution of the CNLC staging of patients diagnosed as liver cancer first from the start of the study to the completion of follow-up | Four years collectively after the study started
The 3-year cumulative incidence of liver cancer in each disease subgroup | Follow up up to 3 years
  The disease types include but are not limited to hepatitis B, hepatitis C, cirrhosis, MAFLD
Early diagnosis rate of HCC in each disease subgroup | Four years collectively after the study started
  The disease types include but are not limited to hepatitis B, hepatitis C, cirrhosis, MAFLD; early diagnosis of HCC is defined as the patient with stage CNLC Ia, Ib and IIa
The compliance rate of each risk group defined at the initial risk stratification | Four years collectively after the study started
  The compliance rates for subjects with very high-risk, high-risk, medium-risk, and low-risk; the compliance rate is defined the same as above

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases , Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China